CLINICAL TRIAL: NCT01752478
Title: Preoperative and Intraoperative Factors Related to the Development of Ptosis After Retinal Surgery
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Other Study IDs: UCSF-Retina
Record Dates: First submitted 2012-12-14; First posted 2012-12-19 (Estimated); Last update posted 2016-05-20 (Estimated); Status verified 2016-05

CONDITIONS: Development of Ptosis After Vitreo-retinal Surgery
Keywords: ptosis; retina surgery; droopy eye lid
MeSH Terms: conditions — Blepharoptosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study to is to determine the incidence of post-operative ptosis in patients undergoing vitreoretinal surgery. An additional purpose is to identify pre-operative and intra-operative factors which correlate to the development of post-operative ptosis in vitreoretinal surgery cases.

DETAILED DESCRIPTION:
This study will evaluate patients who will undergo vitreoretinal surgery at UCSF Medical Center and San Francisco General Hospital. After informed consent has been obtained, the measurement of eyelid parameters such as levator function, palpebral fissure height, upper eyelid crease height, MRD1 and MRD2 will be collected at pre-operative and post-operative follow up visits. External eye photographs taken at each visit will be evaluated by a masked reader who will calculate the eyelid parameters. Dermographic data and intraoperative factors such as operative time and type of procedure will be collected. For statistical analysis, Repeated ANOVA, Paired t-test, Wilcoxon signed rank test, Chi-square test and Pearson's correlation analysis will be calculated with SPSS software.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have vitreoretinal surgery from January 2013

Exclusion Criteria:

* Minors, younger than age 18.
* Patients who have pre-existing ptosis at baseline in the operative eye.
* Patients who are not able to cooperate with eyelid ptosis measurements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient who undergo vitreoretinal surgery at the University of California, San Francisco, and San Francisco General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2013-01; Primary Completion 2016-05 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Reduction of levator function | Baseline to 6 months
  Difference between levator function at baseline and 6 months after surgery

SECONDARY OUTCOMES:
Operative time | At operation
  Record of operative surgical time in each type of operation
Change of palpebral fissure height, MRD1 and MRD2 | Baseline to 6 months
  Difference in palpebral fissure height, MRD1 and MRD2 between baseline and each post-operative visit.
Incidence of ptosis | baseline to 6 months
  Incidence of clinically significant ptosis, defined as upper eyelid drooping of more than 2 mm.

CONTACTS AND LOCATIONS:
Overall Officials: Jay M Stewart, MD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Edmonson BC, Wulc AE. Ptosis evaluation and management. Otolaryngol Clin North Am. 2005 Oct;38(5):921-46. doi: 10.1016/j.otc.2005.08.012. No abstract available. PMID 16214567
- [Background] Bernardino CR, Rubin PA. Ptosis after cataract surgery. Semin Ophthalmol. 2002 Sep-Dec;17(3-4):144-8. doi: 10.1076/soph.17.3.144.14782. PMID 12759843
- [Background] Paris GL, Quickert MH. Disinsertion of the aponeurosis of the levator palpebrae superioris muscle after cataract extraction. Am J Ophthalmol. 1976 Mar;81(3):337-40. doi: 10.1016/0002-9394(76)90250-6. PMID 1258958
- [Background] Kasbekar SA, Wong V, Young J, Stappler T, Durnian JM. Strabismus following retinal detachment repair: a comparison between scleral buckling and vitrectomy procedures. Eye (Lond). 2011 Sep;25(9):1202-6. doi: 10.1038/eye.2011.152. Epub 2011 Jun 24. PMID 21701526
- [Background] Ropo A, Ruusuvaara P, Nikki P. Ptosis following periocular or general anaesthesia in cataract surgery. Acta Ophthalmol (Copenh). 1992 Apr;70(2):262-5. doi: 10.1111/j.1755-3768.1992.tb04134.x. PMID 1609577
- [Background] Donker DL, Paridaens D, Mooy CM, van den Bosch WA. Blepharoptosis and upper eyelid swelling due to lipogranulomatous inflammation caused by silicone oil. Am J Ophthalmol. 2005 Nov;140(5):934-6. doi: 10.1016/j.ajo.2005.05.028. PMID 16310482
- [Background] Quintyn JC, Genevois O, Ranty ML, Retout A. Silicone oil migration in the eyelid after vitrectomy for retinal detachment. Am J Ophthalmol. 2003 Sep;136(3):540-2. doi: 10.1016/s0002-9394(03)00385-4. PMID 12967812